CLINICAL TRIAL: NCT00905242
Title: Impact of Myfortic on GI Prophylaxis in Maintenance Renal Transplant Patients
Brief Title: Impact of Myfortic on Gastrointestinal (GI) Prophylaxis in Maintenance Renal Transplant Patients
Acronym: MPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Paul Bolin, MD, East Carolina University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CERL080A-US41
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Gastrointestinal Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GI medication — Patients on daily dosing were asked to discontinue their GI medication at baseline. Patients on twice daily dosing were asked to reduce GI medication to once a day at baseline and asked to discontinue GI medication at day 30.

SUMMARY:
The purpose of this study is to determine whether maintenance renal transplant patients receiving Myfortic can reduce or discontinue GI prophylaxis medications.

DETAILED DESCRIPTION:
GI prophylaxis is common post kidney transplant and is routinely used in patients receiving a variety of different immunosuppressive regimens. Cellcept and prednisone are often the biggest concern for GI distress and GI ulcers. Routine use of GI prophylaxis medications post-transplant are potentially one mental obstacle to transplant clinicians being fully persuaded of the GI neutral effect of myfortic in the immunosuppressive regimen. Patients receiving myfortic (as part of the conversion in the US02 study) are theoretically at a reduced risk for GI upset and development of GI ulcers. These patients are ideal candidates to discontinue their GI prophylaxis medications while taking myfortic.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the parent study, US02.
* Patients on GI medications.
* Patients currently receiving Myfortic (all dosages are allowed), neoral or tacrolimus with or without corticosteroids as part of their immunosuppressive regimen for at least two weeks.
* Patients with and/or without mild GI complaints (e.g. upper abdominal pain, dyspepsia, anorexia, nausea, vomiting) with or without diarrhea.
* Females of childbearing potential must have a negative pregnancy test prior to the inclusion period. The test should be performed at Baseline visit. If positive, the patient will not be included. Effective contraception must be used during the trial, and for 4 weeks following discontinuation of the study medication.
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion Criteria:

* Evidence of graft rejection or treatment of acute rejection within 14 days prior to Baseline visit.
* Patients who have received an investigational immunosuppressive drug within 4 weeks prior to study entry.
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.
* Patients with thrombocytopenia (<75,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (<4,000/mm3), and/or hemoglobin <9.0g/dL prior to enrollment.
* Presence of clinically significant infection requiring continued therapy, severe diarrhea or active peptic ulcer disease that would interfere with the appropriate conduct of the study.
* Evidence of severe liver disease (incl. abnormal liver profile i.e. AST, ALT or total bilirubin >or= 3 times ULN).
* Abnormal physical or laboratory findings of clinical significance within 2 weeks of inclusion which would interfere with the objectives of the study.
* Evidence of drug and/or alcohol abuse.
* Inability to self-administer the GSRS, GIQLI and PGWBI questionnaires.
* Patients receiving >10mg/day prednisone dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To determine the success (% of patients) in discontinuing GI medications over the 90-day period or also, % of patients able to maintain reduced doses of GI medications over the 90-day period. | 90 days

SECONDARY OUTCOMES:
To evaluate the cost effectiveness of discontinuing GI medications in transplant recipients. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolin, MD, Principal Investigator — East Carolina University
Locations (1):
- Brody School of Medicine at East Carolina University, Greenville, North Carolina, United States